CLINICAL TRIAL: NCT00028275
Title: Pilot Studies of Gamma Interferon Therapy for Chronic Hepatitis C
Brief Title: Gamma Interferon Therapy for Chronic Hepatitis C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 020072; 02-DK-0072
Record Dates: First submitted 2001-12-18; First posted 2001-12-19 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2003-11

CONDITIONS: Chronic Hepatitis C
Keywords: Hepatitis C Virus; Cirrhosis; Antiviral Agents; Viral Resistance; Alpha Interferon; Hepatitis C; Hepatitis
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C; Fibrosis; Hepatitis | interventions — Interferon-gamma

INTERVENTIONS:
Drug: Gamma Interferon 1b

SUMMARY:
This study will test whether gamma interferon is effective in treating chronic hepatitis C infection-a long-lasting viral infection affecting the liver. One-third of patients with hepatitis C infection develop cirrhosis of the liver, which can lead to liver failure or liver cancer. The current treatment for hepatitis C infection is pegylated alpha interferon (peginterferon) plus ribavirin; however, this treatment is successful in only about half of patients. Gamma interferon works similarly to alpha interferon, but through different pathways, and therefore might be helpful in patients who do not respond to alpha interferon.

Patients 18 years of age and older with chronic hepatitis C infection, genotype 1, who did not respond to alpha interferon and ribavirin therapy may be eligible for this study. (Genotype 1 is a strain of hepatitis C virus that has a lower treatment success rate.)

Potential participants will be admitted to the NIH Clinical Center for 2 to 3 days for a medical evaluation to determine eligibility for the study and, if enrolled, to begin gamma interferon therapy. Screening will include a medical history and physical examination, blood and urine tests, and possibly chest X-ray, abdominal ultrasound, and psychiatric evaluation.

Participants will receive injections of gamma interferon under the skin 3 times a week for 4 weeks (a total of 12 injections). They will be randomly assigned to receive either 100 or 200 micrograms of drug per injection. Blood will be drawn just before the first injection and then 6, 12, 24 and 48 hours later to monitor changes in the levels of hepatitis C virus and immune responses to treatment. The amount and rapidity of decrease in virus will be compared with what occurs with alpha interferon treatment to define the relative effectiveness of gamma interferon. (Patients may leave the hospital at any time after the first day, but must return in time for the final blood test.)

Patients will be seen in the clinic each week during treatment to report symptoms and drug side effects and to have blood drawn for routine tests and viral levels. After the 4-week treatment is completed, patients will return for follow-up visits at weeks 6 and 8 for routine blood tests.

DETAILED DESCRIPTION:
We will treat 20 patients with chronic hepatitis C using gamma interferon 1b in doses of either 100 or 200 mcg thrice weekly for four weeks while monitoring them at regular, timed intervals for hepatitis C virus (HCV) RNA levels and immunological responses to HCV antigens. Patients with chronic hepatitis C will be eligible if they have failed to have responded to a previous course of alpha interferon and ribavirin and have raised serum aminotransferase levels, HCV genotype 1 and HCV RNA in serum in levels greater than 10,000 copies/ml. The 20 patients will include 10 patients who were treated and did not become HCV RNA negative during therapy (Group A: non-responders) and 10 who were treated and became HCV RNA negative during therapy but relapsed thereafter (Group B: relapsers). After a medical evaluation and monitoring for HCV RNA levels, patients will be randomized to receive either 100 or 200 mcg of gamma interferon 1b (provided by InterMune Pharmaceuticals, Inc) subcutaneously three times weekly for 4 weeks. Patients will have blood tested for HCV RNA levels at 0, 6, 12, 18, 24, and 48 hours after the initial injection and then weekly during treatment, followed by 2 and 4 weeks thereafter. T cell responses to HCV antigens will be assessed before treatment, after 4 weeks of therapy and again 4 weeks thereafter. Patients will also be monitored for side effects and changes in routine liver tests and complete blood counts.

This is a pilot study in a small number of patients which is aimed at assessing whether gamma interferon has antiviral and immunological effects against hepatitis C, whether these effects appear to be dose related, and whether they are similar in timing and degree to those of alpha interferon. Demonstration of an antiviral effect would lead to more extensive trials in larger numbers of patients, treated for longer periods.

ELIGIBILITY:
INCLUSION CRITERIA:

Age 18 years or above, male or female.

Serum alanine or asparate aminotransferase activities that are above the upper limit of normal (ALT greater than 41 or AST greater than 31 IU/L).

Presence of anti-HCV in serum.

Presence of HCV RNA genotype1 in serum at levels above 10,000 copies/ml.

Previous adequate therapy with alpha interferon and ribavirin without a sustained virological response. An adequate course of therapy is defined as at least 24 weeks of alpha interferon in starting doses of 3 million units thrice weekly and ribavirin in starting doses of at least 1000 mg daily. Patients who initiated therapy at these doses, but required dose modification due to side effects will also be eligible.

Written informed consent.

EXCLUSION CRITERIA:

Decompensated liver disease, as marked by bilirubin greater than 4 mg%, albumin less than 3.0 gm%, prothrombin time greater than 2 sec prolonged, or history of bleeding esophageal varices, ascites or hepatic encephalopathy. Patients with ALT levels greater than 1000 U/L (greater than 25 times ULN) will not be enrolled but may be followed until three determinations are below this level.

Pregnancy, or in women of child-bearing potential or in spouses of such women, inability to practice adequate contraception, defined as vasectomy in men, tubal ligation in women, or use of condoms and spermacide, or birth control pills, or an intrauterine device.

Significant systemic or major illnesses other than liver disease, including congestive heart failure, ischemic heart disease, angina pectoris, cerebrovascular disease, renal failure (creatinine clearance less than 50 ml/min), organ transplantation, serious psychiatric disease or depression.

Pre-existing, severe bone marrow compromise; anemia (hematocrit less than 34%), neutropenia (less than 1000 polymorphonuclear cells/mm(3)) or thrombocytopenia (less than 70,000 cells/mm(3)).

Evidence of another form of liver disease in addition to viral hepatitis (for example autoimmune liver disease, Wilson's disease, alcoholic liver disease, hemochromatosis, alpha-1-antitrypsin deficiency).

Active substance abuse, such as alcohol, inhaled or injection drugs within the previous six months.

Serious autoimmune disease that, in the opinion of the investigators, might be worsened by interferon therapy, such as lupus erythematous, rheumatoid arthritis or Crohn's disease.

Evidence of hepatocellular carcinoma; either alphafetoprotein (AFP) levels greater than 50 ng/ml (normal less than 9 ng/ml) and/or ultrasound (or other imaging study) demonstrating a mass suggestive of liver cancer.

Human immunodeficiency virus infection, as shown by presence of anti-HIV.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 2001-12; Study Completion 2003-11

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK), Bethesda, Maryland, United States

REFERENCES:
- [Background] Liang TJ, Rehermann B, Seeff LB, Hoofnagle JH. Pathogenesis, natural history, treatment, and prevention of hepatitis C. Ann Intern Med. 2000 Feb 15;132(4):296-305. doi: 10.7326/0003-4819-132-4-200002150-00008. PMID 10681285
- [Background] Lauer GM, Walker BD. Hepatitis C virus infection. N Engl J Med. 2001 Jul 5;345(1):41-52. doi: 10.1056/NEJM200107053450107. No abstract available. PMID 11439948
- [Background] Kiyosawa K, Sodeyama T, Tanaka E, Gibo Y, Yoshizawa K, Nakano Y, Furuta S, Akahane Y, Nishioka K, Purcell RH, et al. Interrelationship of blood transfusion, non-A, non-B hepatitis and hepatocellular carcinoma: analysis by detection of antibody to hepatitis C virus. Hepatology. 1990 Oct;12(4 Pt 1):671-5. doi: 10.1002/hep.1840120409. PMID 2170265